CLINICAL TRIAL: NCT07376382
Title: A Randomized, Open-label, Multicenter, Phase III Clinical Trial to Evaluate the Safety and Efficacy of SYS6010 in Combination With Osimertinib in Patients With EGFR-mutant Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Phase Ⅲ Clinical Study of SYS6010 in Combination With Osimertinib in Patients With Locally Advanced or Metastatic NSCLC
Acronym: SYNSTAR-02
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-002
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Multicenter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6010 combination (Experimental): SYS6010 + Osimertinib
  Interventions: Drug: SYS6010; Drug: Osimertinib
- Osimertinib (Active Comparator): Osimertinib
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: SYS6010 — SYS6010，intravenous injection
  Arms: SYS6010 combination
Drug: Osimertinib — Osimertinib 80mg P.O. QD

SUMMARY:
This study is a randomized, open-label, multicenter Phase III clinical trial evaluating patients with EGFR-mutant locally advanced or metastatic NSCLC. The Phase III study is planned to enroll approximately 450 participants, who will be randomized in a 1:1 ratio into the following groups:

Experimental group: SYS6010 + Osimertinib Control group: Osimertinib

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 (inclusive) years old, regardless of gender;
2. Patients with pathologically confirmed locally advanced or metastatic NSCLC, including: patients with stage IIIB or IIIC based on AJCC staging version 8 who are not suitable for surgical resection or radical chemoradiotherapy, or patients with stage IV NSCLC. For the dose escalation phase, patients must have EGFR-mutant locally advanced or metastatic NSCLC that has failed previous standard therapy, and for the dose selection phase and phase III study, patients must have EGFR-mutant locally advanced or metastatic NSCLC, which has not received EGFR-TKIs or other systemic therapy before. Patients who have received adjuvant/neoadjuvant chemotherapy may be included if disease progression occurred at least 6 months after completing treatment;
3. Carry at least one EGFR-sensitive mutation (ex19del or L858R, which can be combined with other EGFR mutations). EGFR mutation: Stage Ib: can be enrolled based on previous test results. Phase III: Take the test results of the central laboratory as the admission group;
4. At least one measurable lesion confirmed by CT or MRI, as defined by RECIST v1.1 criteria;
5. ECOG performance status score 0-1;
6. Expected survival ≥ 3 months;
7. Major organ function meets the relevant laboratory test standards for hematology, renal function, liver function, and coagulation within 7 days prior to treatment;
8. Women of childbearing age had a negative blood pregnancy test within 7 days prior to the first use of study drug. Participants must agree to take effective contraceptive measures from signing the informed consent form to 7 months after the last dose, during which women are non-breastfeeding and men avoid sperm donation;
9. Volunteer to participate in this clinical study, understand the study procedures, and be able to sign a written informed consent form.

Exclusion Criteria:

1. Patients with meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or active CNS metastases;
2. History of other malignant tumors within 3 years prior to the first use of study drug, except for the following conditions: cured skin basal cell or squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, or cervical carcinoma in situ, etc.;
3. Known allergies to SYS6010 or any ingredient of Osimertinib, or to humanized monoclonal antibodies;
4. Adverse events caused by prior anti-tumor therapy that have not resolved to ≤ Grade 1 (as per NCI-CTCAE v6.0), except for Grade 2 alopecia or peripheral neuropathy deemed by the investigator not to pose a safety risk;
5. Use of any of the medications or treatments within the specified washout period (prior to first dose of study drug)
6. History of serious cardiovascular or cerebrovascular conditions within 6 months prior to the first dose, including but not limited to:Severe arrhythmias (e.g., ventricular arrhythmias requiring clinical intervention, third-degree atrioventricular block, QTcF > 470 ms) (Fridericia formula: QTcF = QT/RR0.33, RR = 60/heart rate). Myocardial infarction, unstable angina, aortic dissection, angioplasty, or coronary artery bypass surgery. NYHA class II or higher heart failure with LVEF < 50%.Stroke or other grade ≥ 3 cardiovascular/cerebrovascular events. pulmonary embolism.
7. Patients who have a history of ILD/non-infectious pneumonitis treated with corticosteroids in the past, currently have ILD/non-infectious pneumonitis, for whom imaging examinations at screening cannot rule out ILD/non-infectious pneumonitis, or whose pulmonary function test indicates severe ventilatory dysfunction and/or decreased diffusion capacity;
8. Severe infection within 4 weeks prior to the first dose, such as bacteremia requiring hospitalization, severe pneumonia, or active pulmonary tuberculosis; Active systemic infections requiring antibiotics within 2 weeks prior to administration;
9. Currently suffering from a skin condition requiring oral or vein administration;
10. Participants with active autoimmune disease or a history of autoimmune disease (e.g., ulcerative colitis or Crohn's disease) are excluded from the study. However, participants with the following conditions may be considered eligible for further screening: those with well-controlled type 1 diabetes, well-controlled hypothyroidism requiring only hormone replacement therapy, skin conditions not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia), or diseases unlikely to relapse even when exposed to external triggers;
11. Pleural or peritoneal effusion or pericardial effusion requiring clinical intervention;
12. Conditions that seriously affect gastrointestinal absorption as judged by the investigator (such as Persistent nausea, vomiting, chronic gastrointestinal diseases, gastrointestinal surgery, etc.);
13. Active HBV or HCV infection (hepatitis B surface antigen and/or hepatitis B core antibody positive and HBV DNA copy number ≥ 1 × 104 copy number/mL or ≥ 2000 IU/mL, HCV antibody positive and HCV RNA higher than the lower detection limit of the analytical method), Note: For HBsAg positive, it is recommended to start antiviral therapy before the first use of study drug, and Nucleosides analogs such as Entecavir and Tenofovir disoproxil are recommended);
14. History of immunodeficiency (including positive HIV test, other acquired, congenital immunodeficiency diseases), history of allogeneic stem cell or organ transplantation;
15. Other conditions (e.g. mental illness, macular cystic edema, severe corneal diseases, uncontrolled or poorly controlled hypertension and diabetes, active bleeding, etc.) that the investigator considers inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2026-12-12 (Estimated); Study Completion 2029-06-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) evaluated by IRC | Up to 3.5 years
  PFS is defined as the time from the date of randomization to the first documentation of PD as assessed by investigator per RECIST v.1.1, or death due to any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) evaluated by investigator | Up to 2.5 years
  PFS is defined as the time from the date of randomization to the first documentation of PD as assessed by investigator per RECIST v.1.1, or death due to any cause, whichever occurs earlier.
Overall survival (OS) | Up to 2.5 years
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the participant is known to be alive.
Objective Response Rate (ORR) | Up to 2.5 years
  Objective response rate is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v.1.1.
Duration of Response (DOR) | Up to 2.5 years
  DOR is defined as the time from the date of the first confirmed objective response (CR or PR that is subsequently confirmed) to the date of the first documented disease progression (PD) per RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 2.5 years
  The percentage of participants who experience a best response of CR, PR or stable disease (SD).
Incidence of adverse events | Up to 2.5 years
Incidence of Anti-Drug Antibody (ADA) | Up to 2.5 years
Blood concentration of SYS6010 | Up to 2.5 years